CLINICAL TRIAL: NCT02430415
Title: A Randomized Trial on Comparison of Effects of Two Lightwand Intubation Techniques on Cervical Spine Motion: Laryngoscope-assisted vs. Conventional Lightwand Intubation
Brief Title: Laryngoscope-assisted Lightwand Intubation and Cervical Spine Motion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: LALI
Record Dates: First submitted 2015-04-22; First posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Intubation; Difficult

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): laryngoscope-assisted lightwand intubation - traditional lightwand intubation
  Interventions: Device: laryngoscope-assisted lightwand intubation; Device: traditional lightwand intubation
- Group B (Experimental): traditional lightwand intubation - laryngoscope-assisted lightwand intubation
  Interventions: Device: laryngoscope-assisted lightwand intubation; Device: traditional lightwand intubation

INTERVENTIONS:
Device: laryngoscope-assisted lightwand intubation — laryngoscope-assisted lightwand intubation
Device: traditional lightwand intubation — traditional lightwand intubation

SUMMARY:
The aim of the study is to compare the effect of the laryngoscope-assisted lightwand intubation technique vs. the conventional lightwand intubation technique on the cervical spine motion during intubation in patients with the simulated cervical immobilization.

DETAILED DESCRIPTION:
In clinical practice, the investigators have occasionally experienced some difficulties in the lightwand intubation in patients with cervical spine instability because manual in-line stabilization during intubation hinders free movements of the lightwand such as advancement, withdrawal, and scooping in the oral cavity. For this reason, jaw thrust is often used to secure enough space for free movements of the lightwand in the oral cavity in the traditional lightwand intubation technique. A recent study showed that laryngoscope-assisted lightwand intubation provided more successful intubation on the first attempt and less scooping movement than the traditional lightwand intubation by facilitating free movements of the lightwand in the oral cavity in patients with cervical immobilization during intubation for cervical spine surgery. In the laryngoscope-assisted lightwand intubation technique, the direct laryngoscope may provide sufficient space for free movements of the lightwand in the oral cavity without jaw thrust, which can result in cervical spine movement. However, the effect of the laryngoscope-assisted lightwand intubation technique on cervical spine motion is not investigated yet.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists physical status of 1-2 and age of 18-80 years undergoing elective endovascular coiling to secure cerebral aneurysm under general anesthesia in neuroangiographic rooms.

Exclusion Criteria:

* Patients with the upper airway abnormalities, such as inflammation, abscesses, tumours, polyps, or trauma.
* Patients with past medical history of gastro-oesophageal reflux disease and previous airway surgery, a high risk of aspiration, coagulation disorders, or Hunt Hess grade of 3-5.
* Body mass index > 30

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
maximum cervical spine motion | during tracheal intubation
  maximum angles measured at the occiput-C1, C1-C2, C2-C5 segments.

SECONDARY OUTCOMES:
intubation time | during tracheal intubation
number of intubation trial | during tracheal intubation
sore throat, pain score | after extubation ~ postoperative day 1

CONTACTS AND LOCATIONS:
Overall Officials: Hee Pyung Park, MD PhD, Principal Investigator — Seoul National University of Hospital

REFERENCES:
- [Background] Turkstra TP, Craen RA, Pelz DM, Gelb AW. Cervical spine motion: a fluoroscopic comparison during intubation with lighted stylet, GlideScope, and Macintosh laryngoscope. Anesth Analg. 2005 Sep;101(3):910-915. doi: 10.1213/01.ane.0000166975.38649.27. PMID 16116013
- [Background] Davis L, Cook-Sather SD, Schreiner MS. Lighted stylet tracheal intubation: a review. Anesth Analg. 2000 Mar;90(3):745-56. doi: 10.1097/00000539-200003000-00044. No abstract available. PMID 10702469
- [Derived] Kim TK, Son JD, Seo H, Lee YS, Bae J, Park HP. A Randomized Crossover Study Comparing Cervical Spine Motion During Intubation Between Two Lightwand Intubation Techniques in Patients With Simulated Cervical Immobilization: Laryngoscope-Assisted Versus Conventional Lightwand Intubation. Anesth Analg. 2017 Aug;125(2):485-490. doi: 10.1213/ANE.0000000000001813. PMID 28244946